CLINICAL TRIAL: NCT01901406
Title: Change of Retinally-Induced Aniseikonia in Patients With Epiretinal Membrane After Vitrectomy
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 3-2013-0094
Record Dates: First submitted 2013-07-02; First posted 2013-07-17 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Epiretinal Membranectomy
Keywords: epiretinal membrane, stereopsis, aniseikonia
MeSH Terms: conditions — Epiretinal Membrane; Aniseikonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ERM: idiopathic epiretinal membrane patients

SUMMARY:
Epiretinal membrane is common disease, affecting 5~10 % incidence over 60 years old population. It reduce visual acuity, cause metamorphopsia. In the past, vitrectomy and epiretinal membranectomy was indicated in patients with visual acuity less than 20/40, but nowadays with technical improvement and surgical instrument renovation, it seems to have been changed the surgical indication. Therefore, we plan to evaluate the changes of binocular visual acuity, aniseikonia in patients with epiretinal membrane.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic epiretinal membrane who had impaired vision or metamorphopsia, want to undergo vitrectomy
* Age more than 20 years and less than 90 years old

Exclusion Criteria:

* secondary epiretinal membrane due to retinal surgery,
* impaired visual acuity less than 20/40 in the normal eye(Snellen chart) due to severe cataract
* glaucoma patients
* complication during vitrectomy (ex. Retinal tear, silicone oil injection, …)
* other retinal disease except epiretinal membrane
* other ocular surgery history within 3 months
* intellectual problems or illiterate whom could not obtained informed consent

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with epiretinal membrane who had metamorphopsia or had imparied vision, therefore planned to undergo vitrectomy
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Changes of Stereopsis tested by TNO test (arc of second) | from Initial screening day before surgey to postoperative 6 months
  Stereopsis is normal binocular vision. Its presence or absence is an important indicator of the state of binocularity. The TNO test is graded to provide retinal disparities ranging from 15 to 480 second of arc.
Titmus test (arc of second) | from Initial screening day before surgey to postoperative 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Vision Research, Department of Ophthalmology, Gangnam Severance Hospital, Seoul, South Korea